CLINICAL TRIAL: NCT05609461
Title: Investigation of the Effect of Orthosis Use for Control of Knee Hyperextension in Chronic Stroke Patients by Kinematic Analysis
Brief Title: Investigation of the Effect of Orthosis Use for Control of Knee Hyperextension in Chronic Stroke Patients
Status: Withdrawn | Type: Observational
Why Stopped: Necessary equipment could not be provided.
Sponsor: Hacettepe University (Other)
Collaborators: Atılım University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: E-59394181-604.01.02-47710
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: Gait Analysis; Foot-Ankle Orthosis; Knee Hyperextension; Kinematic Analysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic stroke patients with knee hyperextension

SUMMARY:
The aim of this study is to examine the effect of using foot-ankle orthosis at different angles on hyperextension control in stroke patients.

The hypotheses of the study are:

Hypothesis 1:

Ho: The foot-ankle orthosis, which fixes the ankle at different angles (3 degrees of dorsiflexion - 5 degrees of dorsiflexion) in stroke patients, has no effect on the control of knee hyperextension.

H1: Foot-ankle orthosis, which fixes the ankle at different angles (3 degrees of dorsiflexion - 5 degrees of dorsiflexion) in stroke patients, has an effect on the control of knee hyperextension.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40 and 65
* Six months must have passed since the stroke.
* Ambulation regardless of the use of a walking aid (walker, cane, or tripod)
* Obtaining between 0 and 3 Modified Rankin Score points
* A score of 24 or higher on the Mini Mental Test is required to pass.
* Hyperextension during the stance phase of gait.
* Participating voluntarily in the study

Exclusion Criteria:

* Having a history of more than one stroke
* Dementia is known to exist
* Having a diagnosed orthopedic, mental, or neurological condition
* Having a circumstance that impedes communication
* Having a history of lower extremity and gait-related surgeries

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Patients with Knee Hyperextension
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Kinematic Analysis | Baseline
  At the specified anatomical sites of the participants, reflective signs will be placed. The participants will be required to walk 5 meters. The three-dimensional positions of these reflective marks will be captured by the 8-camera Vicon motion capture system. Using the blade software, it will be moved to the computer environment and kinematic data will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Armutlu, Prof. Dr., Study Chair — Hacettepe University; Süleyman Korkusuz, MSc, Principal Investigator — Hacettepe University; Sibel Kibar, Assoc. Prof., Study Chair — Atılım University; Serdar Arıtan, Asst.Prof, Study Chair — Hacettepe University; Nihat Özgören, MSc, Study Chair — Hacettepe University; Büşra Seçkinoğulları, Msc, Study Chair — Hacettepe University; Ayla Fil Balkan, Assoc.Prof, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geerars M, Minnaar-van der Feen N, Huisstede BMA. Treatment of knee hyperextension in post-stroke gait. A systematic review. Gait Posture. 2022 Jan;91:137-148. doi: 10.1016/j.gaitpost.2021.08.016. Epub 2021 Aug 24. PMID 34695721
- [Background] Bae DY, Shin JH, Kim JS. Effects of dorsiflexor functional electrical stimulation compared to an ankle/foot orthosis on stroke-related genu recurvatum gait. J Phys Ther Sci. 2019 Nov;31(11):865-868. doi: 10.1589/jpts.31.865. Epub 2019 Nov 26. PMID 31871367
- [Background] Kobayashi T, Orendurff MS, Singer ML, Gao F, Daly WK, Foreman KB. Reduction of genu recurvatum through adjustment of plantarflexion resistance of an articulated ankle-foot orthosis in individuals post-stroke. Clin Biomech (Bristol). 2016 Jun;35:81-5. doi: 10.1016/j.clinbiomech.2016.04.011. Epub 2016 Apr 23. PMID 27136122